CLINICAL TRIAL: NCT07034794
Title: A Randomized, Triple-blind, Placebo Controlled, Parallel Clinical Trial to Examine Lysoveta on Cognitive Function in Healthy Adults With Self-perceived Memory Problems
Brief Title: A Clinical Trial to Examine Lysoveta on Cognitive Function in Healthy Adults With Self-perceived Memory Problems
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aker BioMarine Human Ingredients AS (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25AKCFA01
Record Dates: First submitted 2025-06-12; First posted 2025-06-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-06

CONDITIONS: Healthy; Memory Problems
Keywords: Lysoveta; Memory Problems; Hydrolyzed krill oil
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lysoveta (Experimental): This group receives 3 capsules containing 500 mg/capsule of Lysoveta, a hydrolyzed krill oil rich in omega-3 fatty acid bound to lysophosphatidylcholine.
  Interventions: Dietary Supplement: Lysoveta
- Placebo (Placebo Comparator): This group receives medium-chain triglyceride (MCT) oil, maize oil, olive oil, and palm kernel oil daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lysoveta — The Lysoveta capsules contain 500 mg of lysophosphatidylcholine-rich oil extract of Antarctic krill.
  Arms: Lysoveta
Other: Placebo — The placebo capsules contain medium-chain triglyceride (MCT) oil, maize oil, olive oil, and palm kernel oil.
  Arms: Placebo

SUMMARY:
The study is a randomized, placebo-controlled, triple-blind, parallel group trial, in which the effect of krill oil is investigated in healthy volunteers with self-perceived memory problems. Volunteers are randomly allocated to the 2 study groups including placebo and Lysoveta. Over the whole study period, volunteers will be asked to complete questionnaires to evaluate cognitive performance and mood throughout the duration of the trial.

The goal of this clinical trial is to examine Lysoveta on cognitive function in healthy adults with self-perceived memory problems. The main question it aims to answer is:

What is the difference in change in episodic, working and spatial memory as assessed by the Computerized Mental Performance Assessment System (COMPASS) between Lysoveta and placebo?

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 50 and 75 years, inclusive
2. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle and agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence and agrees to use contraception if planning on becoming sexually active during the study
3. Self-reported memory problems as assessed by a combined score of ≥ 6 on Everyday Memory Questionnaire (EMQ) questions 1, 2 and 18 at screening
4. Agrees to avoid moderate-vigorous exercise 12 hours prior to post-screening clinic visits
5. Agrees to avoid high sources of caffeine (e.g., supplements, tea, coffee, energy drinks), NSAIDs, and alcohol consumption for 24 hours prior to post-screening clinic visits
6. Agrees to avoid first generation anti-allergy medication for 48 hours prior to post-screening clinic visits
7. Agrees to maintain current lifestyle habits (diet, physical activity, medications, supplements, and sleep) as much as possible throughout the study
8. Agrees to avoid travelling between two or more time zones within one week of in-clinic visits
9. Willingness to complete questionnaires, records and diaries associated with the study and to complete all clinic visits
10. Provided voluntary, written, informed consent to participate in the study
11. Healthy as determined by medical history and laboratory results as assessed by Qualified Investigator (QI)

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance preventing consumption of investigational product or placebo ingredients, including seafood and/or shellfish
3. Dementia or other significant cognitive impairment as assessed by the Mini Mental State Exam-2 Standard Version (MMSE-2) with a score < 24 at screening
4. Self-reported confirmation of any significant neuropsychological condition and/or cognitive impairment (e.g., Schizophrenia, bipolar disorder, post-traumatic stress disorder, brain injury, neurodegenerative disease, infections, insomnia, depression, epileptic or other seizure-related disorders) that could interfere with study participation as assessed by the QI
5. Regularly consumes two or more servings of fatty fish per week as assessed by the QI
6. Self-reported color blindness/weakness as assessed by the QI
7. Current employment that calls for overnight shiftwork as assessed by the QI
8. Postmenopausal confusion, as assessed by the QI
9. Unstable metabolic disease or chronic diseases as assessed by the QI
10. Current or history of any significant diseases of the gastrointestinal tract as assessed by the QI
11. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI (See Section 7.3)
12. Type I diabetes
13. Type II diabetes if on insulin treatment. Type II diabetics on stable medication for at least three months and an HbA1c of <8.0% may be included after assessment by the QI on a case-by-case basis
14. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
15. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
16. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
17. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
18. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
19. Individuals with an autoimmune disease or are immune compromised as assessed by the QI
20. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis as assessed by the QI
21. Self-reported confirmation of blood/bleeding disorders as assessed by the QI
22. Use of medical cannabinoid products
23. Chronic use of cannabinoid products (>2 times/week). Occasional users will be required to washout and abstain for the duration of the study period
24. Irregular use of tobacco or nicotine products in the past one month, as assessed by the QI
25. Alcohol intake average of >2 standard drinks per day as assessed by the QI
26. Alcohol or drug abuse within the last 12 months
27. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy or safety of the investigational product (Section 7.3)
28. Clinically significant abnormal laboratory results at screening as assessed by the QI
29. Blood donation 30 days prior to baseline, during the study, or a planned donation within 30 days of the last study visit
30. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
31. Individuals who are unable to give informed consent
32. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-12-06 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The difference in change in episodic, working and spatial memory | Day 0 (baseline) to 112
  The difference in change in episodic, working and spatial memory as assessed by the Computerized Mental Performance Assessment System (COMPASS) from baseline at Day 112 between Lysoveta and placebo. COMPASS delivers randomly generated tasks for each participant that are selected from a wide range of pre-programmed standard cognitive tests based on the objective of the study.

SECONDARY OUTCOMES:
The difference in the change in episodic, working and spatial memory | Day 0 to 14
  The difference in the change from baseline between Lysoveta and placebo in Episodic, working and spatial memory as assessed by COMPASS at Day 14. COMPASS delivers randomly generated tasks for each participant that are selected from a wide range of pre-programmed standard cognitive tests based on the objective of the study.
The difference in the change in executive function | Day 0 to 14
  The difference in the change from baseline between Lysoveta and placebo in executive function as assessed by COMPASS at Days 14. COMPASS delivers randomly generated tasks for each participant that are selected from a wide range of pre-programmed standard cognitive tests based on the objective of the study.
The difference in the change in executive function | Day 0 to 112
  The difference in the change from baseline between Lysoveta and placebo in executive function as assessed by COMPASS at Days 112. COMPASS delivers randomly generated tasks for each participant that are selected from a wide range of pre-programmed standard cognitive tests based on the objective of the study.
The difference in the change in reaction time | Day 0 to 14
  The difference in the change from baseline between Lysoveta and placebo in reaction time as assessed by COMPASS at Days 14. COMPASS delivers randomly generated tasks for each participant that are selected from a wide range of pre-programmed standard cognitive tests based on the objective of the study.
The difference in the change in memory | Day 0 to 112
  The difference in the change from baseline between Lysoveta and placebo in memory as assessed by the Everyday Memory Questionnaire at Day 112. On a 5-point scale: 0 = never, 1 = less than once a week, 2 = once or twice a week, 3 = about once each day, 4 = several times in a day.
The difference in the change in mood | Day 0 to 14
  The difference in the change from baseline between Lysoveta and placebo in mood as assessed by the Profile of Mood States (POMS) at Days 14. POMS is a self-reported assessment of mood that is adaptable to capturing transient and fluctuating feelings, or relatively enduring affect states and contributes to a comprehensive assessment by providing indications of potential mood disturbance. On a scale of "not at all" to "extremely".
The difference in the change in mood | Day 0 to 112
  The difference in the change from baseline between Lysoveta and placebo in mood as assessed by the Profile of Mood States (POMS) at Days 14. POMS is a self-reported assessment of mood that is adaptable to capturing transient and fluctuating feelings, or relatively enduring affect states and contributes to a comprehensive assessment by providing indications of potential mood disturbance. On a scale of "not at all" to "extremely".
The difference in the change in omega-3 status | Day 0 to 56
  The difference in the change from baseline between Lysoveta and placebo in omega-3 status as assessed by the Omega-3 Index (omega-3 blood concentration) at Days 56.
The difference in the change in omega-3 status | Day 0 to 112
  The difference in the change from baseline between Lysoveta and placebo in omega-3 status as assessed by the Omega-3 Index (omega-3 blood concentration) at Days 112.
The difference in the change in serum brain-derived neurotrophic factor (BDNF) | Day 0 to 56
  The difference in the change from baseline between Lysoveta and placebo in serum brain-derived neurotrophic factor (BDNF) at Day 56
The difference in the change in serum brain-derived neurotrophic factor (BDNF) | Day 0 to 112
  The difference in the change from baseline between Lysoveta and placebo in serum brain-derived neurotrophic factor (BDNF) at Day 112

OTHER OUTCOMES:
Incidence of post-emergent adverse events (AE) | Day 0 to 112
  Incidence of post-emergent adverse events (AE)
Clinically relevant changes in blood pressure after supplementation | Day 0 to 112
  Clinically relevant changes in blood pressure after supplementation
Clinically relevant changes in heart rate after supplementation | Day 0 to 112
  Clinically relevant changes in heart rate after supplementation
Clinically relevant changes in clinical chemistry | Day 0 to 112
  Clinically relevant changes in aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) after supplementation
Clinically relevant changes in clinical chemistry | Day 0 to 112
  Clinically relevant changes in total bilirubin after supplementation
Clinically relevant changes in clinical chemistry | Day 0 to 112
  Clinically relevant changes in creatinine after supplementation
Clinically relevant changes in clinical chemistry | Day 0 to 112
  Clinically relevant changes in estimated glomerular filtration rate (eGFR) after supplementation
Clinically relevant changes in clinical chemistry | Day 0 to 112
  Clinically relevant changes in glucose after supplementation
Clinically relevant changes in complete blood count after supplementation | Day 0 to 112
  Clinically relevant changes in complete blood count after supplementation
Clinically relevant changes in lipid profile after supplementation | Day 0 to 112
  Clinically relevant changes in triglycerides (TG) after supplementation
Clinically relevant changes in lipid profile after supplementation | Day 0 to 112
  Clinically relevant changes in total cholesterol (TC) after supplementation
Clinically relevant changes in lipid profile after supplementation | Day 0 to 112
  Clinically relevant changes in high-density lipoprotein cholesterol (HDL-C) after supplementation
Clinically relevant changes in lipid profile after supplementation | Day 0 to 112
  Clinically relevant changes in non-HDL-C after supplementation
Clinically relevant changes in lipid profile after supplementation | Day 0 to 112
  Clinically relevant changes in low-density lipoprotein cholesterol (LDL-C), (TC:HDL-C, TG:HDL-C, and LDL-C:HDL-C ratios) after supplementation
Clinically relevant changes in lipid profile after supplementation | Day 0 to 112
  Clinically relevant changes in oxidized LDL (oxLDL)* after supplementation
Inflammatory markers as assessed by C-reactive protein (CRP) | Day 0 to 112
  Inflammatory markers as assessed by C-reactive protein (CRP)
The difference in change in LPC-DHA and LPC-EPA | Day 14 to 112
  The difference in change in LPC-DHA and LPC-EPA from baseline at Days 14 and 112
The difference in change in biological age, as assessed by epigenetic analysis | Day 0 to 112
  The difference in change in biological age, as assessed by epigenetic analysis at baseline and Day 112

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada